CLINICAL TRIAL: NCT01866475
Title: A Study to Determine the Safety of Continuous Intraosseous Vascular Access Over a Period of 48 Hours
Brief Title: Continuous Intraosseous Vascular Access Over 48 Hours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vidacare Corporation (Industry)
Responsible Party: Sponsor
Organization: Teleflex (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2011-16
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Results first posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Intraosseous Vascular Access
Keywords: IO access; Intraosseous vascular access; EZ-IO

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Renal Disease (Active Comparator): Those with mild to moderate renal disease and had an EZ-IO for 48 hours
  Interventions: Device: EZ-IO
- Diabetes (Active Comparator): Those with controlled diabetes and had an EZ-IO for 48 hours
  Interventions: Device: EZ-IO
- Renal disease and diabetes (Active Comparator): Those with both mild to moderate renal disease and controlled diabetes and had an EZ-IO for 48 hours
  Interventions: Device: EZ-IO
- Healthy adults (Active Comparator): Those who are healthy, defined as lacking co-morbidities that are a study exclusion, and had an EZ-IO for 48 hours
  Interventions: Device: EZ-IO

INTERVENTIONS:
Device: EZ-IO — To have an EZ-IO placed up to 48 hours

SUMMARY:
A prospective study to determine the safety of intraosseous (IO) access for a period up to 48 hours in healthy adult volunteers and volunteers with a history of mild to moderate renal disease and/or controlled diabetes.

DETAILED DESCRIPTION:
A prospective, study to determine the safety of intraosseous (IO) access for a period up to 48 hours, in healthy adult volunteers and volunteers with a history of being health-compromised, including patients with mild to moderate renal disease (National Health and Nutrition Examination Survey Stage 1 to 3) and/or patients with controlled diabetes. Subjects will be randomized to receive IO access in the proximal tibia insertion site or the proximal humerus insertion site using the EZ-IO intraosseous vascular access system. The hypothesis is that there will be no serious complications for the subjects during a 48 hour IO catheter dwell time in either place.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older
* Self Identifying as having poor vascular access
* Healthy or Having at least one of the following conditions:
* Controlled diabetes, as evidenced by a glycosylated hemoglobin A1c (HbA1c) value of less than or equal to 8% at the time of screening. or
* Renal disease, Stages 1 to 3, as evidenced by the presence of albuminuria at the time of screening. Subjects albumin-creatinine ratio (ACR) must fall within the microalbuminuria or macroalbuminuria values: Microalbuminuria - ACR 17-250 mcg/mg for men; 25-355 mcg/mg for women or, Macroalbuminuria- ACR >250 mcg/mg for men; >355 mcg/mg for women

Exclusion Criteria:

* Imprisoned
* Self identifying as pregnant
* Cognitively impaired
* Fracture in target bone
* Excessive tissue and/or absence of adequated anatomical landmarks in target bone
* Signs and symptoms of infection in target area
* IO insertion in past 48 hours, prosthetic limb or joint or other significant orthopedic procedure in target bone
* Intravenous infusion within the past 30 days
* Current use of anti-coagulants
* Previous adverse reaction or known allergy to Lidocaine
* Current cardiac condition requiring pacemaker
* Currently taking beta blockers or calcium channel blockers for heart arrhythmia (use of beta blockers or calcium channel blocker for hypertension is allowed when indication of hypertension can be confirmed by physician
* Previous surgery for peripheral arterial disease
* History of ulcers to the extremities
* History of bilateral lymph node dissection in the arms or legs
* Known sickle-cell disease
* signs or symptoms of vascular disease or vascular insufficiencies to the extremities, as identified upon physical examination
* History of peripheral vascular disease
* Hyperkalemia as evidenced by potassium level greater than 5.1 mmol/L the upper limit of hte normal reference range at screening

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel DeNoia, MD, Principal Investigator — ICON Early Phase Services
Locations (1):
- ICON Early Phase Services, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: November 2014 - January 2016: subjects with controlled diabetes and/or mild renal disease only were enrolled.
  January 2016 - July 2016: healthy subjects and subjects with controlled diabetes and/or mild renal disease were enrolled. Amendment for healthy subjects approved by FDA in advance of implementation.
Period: Overall Study
Arm/Group | Renal Disease | Diabetes | Renal Disease and Diabetes | Healthy Adults
Started | 0 | 40 | 3 | 84
Completed (Completed through day 3 procedures) | 0 | 39 | 3 | 79
Not Completed | 0 | 1 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Four subsets of subjects were targeted for enrollment in the study; those with renal disease, diabetes, renal disease and diabetes, and healthy adults. There were 0 renal disease subjects enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Renal Disease | Diabetes | Renal Disease and Diabetes | Healthy Adults | Total
Number analyzed (Participants) | 0 | 40 | 3 | 84 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 53.6 (11.7) | 47 (12.3) | 41.4 (12.7) | 45.4 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 14 | 1 | 31 | 46
  Male |  | 26 | 2 | 53 | 81
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black |  | 10 | 0 | 17 | 27
  Race/Ethnicity: White |  | 12 | 1 | 41 | 54
  Race/Ethnicity: Asian |  | 0 | 0 | 1 | 1
  Race/Ethnicity: American Indian / Alaska Native |  | 0 | 0 | 1 | 1
  Race/Ethnicity: Native Hawaii / Pacific Islander |  | 0 | 0 | 0 | 0
  Race/Ethnicity: Hispanic / Latino |  | 0 | 0 | 2 | 2
  Race/Ethnicity: White and Hispanic / Latino |  | 17 | 2 | 22 | 41
  Race/Ethnicity: Black and Hispanic / Latino |  | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 40 | 3 | 84 | 127

OUTCOME MEASURES:

1. Primary Outcome: Serious Complications From Intraosseous (IO) Access
Description: Presence of serious complications from 48 hour intraosseous (IO) vascular access using EZ-IO.
Time Frame: 48 hours
Population: Evaluable subjects included in primary endpoint analysis. Non-evaluable subjects, defined by protocol as subjects who withdrew consent or were discontinued from the study for non-compliance or unwillingness to comply with study requirements before completing Day 3 procedures (48 hour dwell time), were replaced. There were 6 non-evaluable subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Disease | Diabetes | Renal Disease and Diabetes | Healthy Adults
Number analyzed (Participants) | 0 | 39 | 3 | 79
Participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Diabetes vs Renal Disease and Diabetes vs Healthy Adults; Test type: Non-Inferiority — This study is designed to test the hypothesis that the IO device has no greater than a 4 percent infection rate. Equivalently, we define success as having at least a 96 percent infection free 48-hour placement; The historical data for the device suggests an infection rate of 0.6 percent per 48 hours or a success rate of 99.4 percent. The formal objective in the design is to reject the one-sided null hypothesis that the success rate is no higher than 96 percent. The analysis will use the exact binomial test and will tolerate a Type I Error rate of 0.05 or less. If we assume a 99.4 percent success rate, the study will have 84 percent power with a sample size of 117 to reject the null hypothesis. If the null hypothesis is rejected, we conclude that the infection rate is less than 4 percent

ADVERSE EVENTS:
Time Frame: 48 hours
Description: Subjects were routinely assessed for adverse events following intraosseous (IO) insertion catheter every 15 minutes for the first 2 hours, then every 2 hours for the remaining 48 hour dwell time. A laboratory test was done at the time of IO catheter removal to assess for osteomyelitis.
  No subjects were enrolled into the Renal Disease arm of the study, therefore the number of participants at risk for Other Adverse Events, All-Cause Mortality, and Serious Adverse Events for this group is zero.
Arm/Group | Renal Disease | Diabetes | Renal Disease and Diabetes | Healthy Adults
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/40 | 0/3 | 0/84
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/40 | 0/3 | 0/84
Other Adverse Events (participants affected / at risk) | 0/0 | 33/40 | 2/3 | 77/84
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Disease (N=0) | Diabetes (N=40) | Renal Disease and Diabetes (N=3) | Healthy Adults (N=84)
Elevated White Blood Cells (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — elevated white blood cells and elevated neutrophils
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Imprint EZ-IO (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Imprint of EZ-IO catheter hub on the skin surface
pain (Surgical and medical procedures) | 0 (0) | 26 (50) | 2 (4) | 75 (76) — pain, without other symptoms, is a known and expected adverse event associated with intraosseous access and infusion
pain - referred pain, distal tibia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Referred pain to distal tibia from right IO site
Scar (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — scar matches demarcation of device hub, hypopigmented at insertion sites
soreness - arm left (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
swelling - IO site (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 5 (5)
Vasovagal response (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
pain- left heel foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
soreness- left knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pain - various focus points (General disorders) | 0 (0) | 7 (7) | 0 (0) | 9 (9)
Skin - local allergy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — superficial phlebitis
burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — left arm, 1st degree burn
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
emesis / nausea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
erythema - knee (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fractured tooth (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
headache (General disorders) | 0 (0) | 7 (10) | 2 (2) | 10 (11)
hoarseness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
junctional heart rate (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
light headedness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
nausea / upset stomach (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 4 (4)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
sinus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
swelling - knee posterior (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No